CLINICAL TRIAL: NCT01675102
Title: Allogeneic HSCT in 17p- CLL in First or Second Partial or Complete Remission at Transplant: a Non-interventional Prospective Study.
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) in 17p- Chronic Lymphocytic Leukemia (CLL)
Acronym: 17p-CLL
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: European Research Initiative on CLL (Unknown)
Responsible Party: Sponsor
Other Study IDs: EBMT-42204420
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: CLL
Keywords: del 17p; chronic lymphocytic leukemia; cll; mutation; p53
MeSH Terms: conditions — Chromosome 17 deletion; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
17p-/p53-mutated chronic lymphocytic leukemia (CLL) is an orphan disease, accounting for approximately 5% of newly diagnosed CLL. This subgroup of patients has a very poor outcome after chemoimmunotherapy. Allogeneic HCT may change the poor prognosis. In a retrospective EBMT-analysis on 44 patients with advanced 17p-CLL 2-year progression-free survival was 45% (95% CI, 30% to 60%) after allogeneic HCT (Allogeneic hematopoietic stem-cell transplantation for chronic lymphocytic leukemia with 17p deletion: a retrospective European Group for Blood and Marrow Transplantation analysis. J Clin Oncol, 2008, 26, 5094-5100).

Referring to these favorable results and small additional series, patients with 17p-CLL requiring therapy are considered to have an indication for allogeneic transplantation by many CLL study groups. Several CLL study groups recommend allogeneic HCT in 17p-CLL as part of the first- or second line treatment.

The aim is to collect additional evidence on allogeneic HCT in 17p-/p53-mutated CLL in first or second remission by a non-interventional prospective study. Patients shall be registered prior to HCT at the Leiden Office in order to rule out a reporting bias after transplantation.

DETAILED DESCRIPTION:
Objective:

The aim is to determine early PFS after allogeneic HCT in first or second remission of 17p-/p53-mutated CLL within an epidemiologic study.

Methods:

Neither the decision for allogeneic transplantation nor specific treatment recommendations for patients with 17p-/p53-mutated CLL are part of the study. Instead, the study protocol refers to EBMT guidelines. Indications for allogeneic stem cell transplantation in chronic lymphocytic leukemia: the EBMT transplant consensus. Leukemia 21, 2007, 12-17). Minimal essential data (MED) A and B, defined by the EBMT, will be collected (www.ebmt.org).

The rate of progression-free survival (PFS) at 1 year after HSCT was selected as primary endpoint. Death, clinical relapse or progression but not immune manipulations (taper of immunosuppression, DLI, rituximab) are considered as treatment failure for PFS. Patients without information on one-year follow up will be considered as having experienced treatment failure. The rate of PFS at 1 year will be calculated by dividing the number of patients without treatment failure by the number of patients who met all selection criteria.

For the calculation of the sample size a fixed sample design was selected. The null hypothesis is that the success-rate for PFS is equal or less than 50%. Referring to the retrospective EBMT survey, PFS at one year after allogeneic HCT is expected to be 70%. According to Fleming-A'Hern (1982) the null hypothesis can be rejected with a power of 80% and an alpha error of 5% if a minimum of 24 out of 37 informative patients did not experience treatment failure during the first year after allogeneic HCT (Machin et al, Sample Size Tables for Clinical Studies, Wiley-Blackwell, 3rd edition, 2009). Taking into account a 10% drop-out rate by violation of inclusion criteria the target number of patients to be included was set at 41 patients.

ELIGIBILITY:
Inclusion Criteria:

* 17p-/p53-mutated CLL by FISH or sequencing, confirmed by review by an experienced laboratory
* first or second partial remission or complete remission at HCT according to the updated NCI-criteria (Hallek 2008)
* MRD diagnostic as part of the local standard follow up
* allogeneic HCT from a matched related or unrelated donor with up to one mismatch refering to HLA-A, -B, -C and DRB1

Exclusion Criteria:

* ex vivo T-cell depletion
* in vivo T-cell depletion with alemtuzumab

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: eligible patients from EBMT centres
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-08-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | 1 year after HSCT

SECONDARY OUTCOMES:
Rate of MRD-negative complete remissions | 1 year after HSCT
Overall survival, cumulative incidence of relapse and non-relapse mortality | 1 year after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schetelig, MD, Principal Investigator — Medizinische Klinik und Poliklinik I, University Hospital Dresden, Germany; Nicolaus Kroeger, MD, Study Chair — BMT Centre, University Hospital Eppendorf, Hamburg, Germany
Locations (10):
- Rigshospitalitet, Copenhagen, Denmark
- University Central Hospital, Helsinki, Finland
- Germany (4):
  - Universitaetsklinikum, Dresden
  - University Hospital Eppendorf, Hamburg
  - University of Heidelberg, Heidelberg
  - Klinik fuer Innere Medzin III, Ulm
- Chaim Sheba Medical Centre, Tel Litwinsky, Israel
- University Hospital, Maastricht, Netherlands
- University Hospital, Lund, Sweden
- City Hospital, Nottingham, United Kingdom